CLINICAL TRIAL: NCT03070717
Title: High Myopia: Extended and Longterm Observation of Pathologic Myopia Patients With the Risk for Developing a Myopic Choroidal Neovascularization (CNV)
Acronym: HELP
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002FDE01
Record Dates: First submitted 2016-02-17; First posted 2017-03-03 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Pathologic Myopia
Keywords: High myopia, shortsightedness, retinal changes
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: Patients with diagnosis of high myopia secondary to an anterior-posterior elongation of the bulbus confirmed by ocular examination in either eye using specific criteria.
  Interventions: Procedure: Observation & Diagnosis

INTERVENTIONS:
Procedure: Observation & Diagnosis — SD-OCT, fundus autofluorescence, fundus photography, optional microperimetry, ophthalmic exams (BCVA, optical biometry), blood sampling.

SUMMARY:
This research project intends to observe patients with high myopia who show pathological retinal changes, in order to evaluate more data on the risk factors for developing mCNV within this research project population in Germany.

ELIGIBILITY:
Inclusion Criteria:

* Male or female caucasian patients ≥ 18 years of age
* Diagnosis of high myopia secondary to an anterior-posterior elongation of the bulbus confirmed by ocular examination in either eye using the following criteria:

  * Ocular ultrasonography or biometry demonstrating anterior-posterior elongation measurement ≥ 26 mm
  * abnormal change in retinal tissue by SD-OCT that are attributed to be caused by high myopia as shown in Table 4-2 of the protocol in the investigator's discretion confirmed by the reading centre

Exclusion Criteria:

* Patients with Diabetes mellitus of any grade
* Patients showing signs of Age-Related Macular Degeneration (AMD), e.g. drusen, characteristic changes in fundus (with shaping or extension of hemorrhages, fibrosis, exudative areas) in either eye
* Acute neovascularization (CNV or iris neovascularization) and intra- or subretinal fluid in either eye at the time of enrolment.
* History of inactive CNV in study eye. Inactive CNV of fellow eye is allowed if treatment was performed more than 12 months before enrolment.
* Any anti vascular endothelial growth factor' (anti-VEGF) or Verteporfin treatment in study eye and anti-VEGF or Verteporfin treatment less than 12 months before enrolment in fellow eye
* History of systemic anti vascular endothelial growth factor' (anti-VEGF) therapy
* Cataract that would prevent an accurate measurement of the axial length of the study eye

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Caucasian adults with high myopia in Germany, recruited on an outpatient basis.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2014-06-12 (Actual); Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Change in retinal morphology by SD-OCT | Baseline, first year, 2nd year, 3rd year
  To exploratively determine the pathogenesis within the project population by assessing and evaluating the risk factors of myopic CNV by measuring the change in retinal morphology with spectral domain optical coherence tomography (SD-OCT).
  Risk factors are defined as choroidal thinning < 50μm, choroidal curvature length > 6300 μm (nasal temporal), lacquer cracks, patchy atrophy > 5mm² and preexisting myopic CNV in second eye.

SECONDARY OUTCOMES:
Change in retinal morphology by fundus autofluorescence | Baseline, first year, 2nd year, 3rd year
  To exploratively determine the pathogenesis within the project population by assessing and evaluating the risk factors of myopic CNV within the project population by measuring the change in retinal morphology with fundus autofluorescence.
  Risk factors are defined as choroidal thinning < 50μm, choroidal curvature length > 6300 μm (nasal temporal), lacquer cracks, patchy atrophy > 5mm² and preexisting myopic CNV in second eye.
Change in retinal morphology by fundus photography | Baseline, first year, 2nd year, 3rd year
  To exploratively determine the pathogenesis within the project population by assessing and evaluating the risk factors of myopic CNV within the project population by measuring the change in retinal morphology with fundus photography.
  Risk factors are defined as choroidal thinning < 50μm, choroidal curvature length > 6300 μm (nasal temporal), lacquer cracks, patchy atrophy > 5mm² and preexisting myopic CNV in second eye.
Change in Best Corrected Visual Acuity (BCVA) by vision testing (Landolt chart or equivalent) | Baseline, 3rd year
  To exploratively determine the pathogenesis within the project population and within the individual patient by change of BCVA from baseline to 3rd year.
Change in refraction error by autorefractometer | Baseline, 3rd year
  To exploratively determine the pathogenesis within the project population and within the individual patient by change of refraction error from baseline to 3rd year.

OTHER OUTCOMES:
Occurence of myopic CNV at the investigator's discretion | From baseline until the date of occurence of myopic CNV at the investigator's discretion (if any), assessed up to 3 years.
  To assess if myopic CNV in study eye and/or fellow eye occured from baseline to 3rd year.
Change in health related quality of life (QoL) by NEI-VFQ-25 questionnaire | Baseline and 3rd year (or at the date of occurence of myopic CNV at the investigator's discretion, if any, whichever comes first, assessed up to 3 years).
  To assess the change in health related QoL by patient reported outcome with the VFQ-25 questionnaire.
Assessment of biomarkers by analyzing blood samples | Baseline and at the date of occurence of myopic CNV at the investigator's discretion, if any, assessed up to 3 years.
  To assess biomarkers which are possibly related to mCNV development. Blood samples will be taken at baseline from all patients who gave separate informed consents. A second sample will only be taken at CNV occurence (if any), assessed up to 3 years. Inflammatory and angiogenic markers will be measured and checked for the potential association to CNV formation.
Assessment of genetic factors by analyzing blood samples | Baseline and at the date of occurence of myopic CNV at the investigator's discretion, if any, assessed up to 3 years.
  To assess genetic factors which are possibly related to mCNV development. Blood samples will be taken at baseline from all patients who gave separate informed consents. A second sample will only be taken at CNV occurence (if any), assessed up to 3 years. Inflammatory and angiogenic markers will be measured and checked for the potential association to CNV formation.
Change in axial length of the bulbus by optical biometry | Baseline, first year, 2nd year, 3rd year
  To assess the change in axial length of the bulbus in both eyes by optical biometry.

CONTACTS AND LOCATIONS:
Locations (22):
- Germany (22):
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Ansbach
  - Novartis Investigative Site, Bad Rothenfelde
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hösbach
  - Novartis Investigative Site, Karlsruhe
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Würzburg

REFERENCES:
- See also: Sponsor website — http://klinischeforschung.novartis.de/doctor/studie-fuer-patienten-mit-starker-kurzsichtigkeit-crfb002fde01/